CLINICAL TRIAL: NCT04650516
Title: Evaluation of Pain Relief in Patients Experiencing Endometriosis-related Pain and Treated With Endocare®
Brief Title: Endocare® (Single Care) in Pain-related Endometriosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lucine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20206-A01541-38
Record Dates: First submitted 2020-11-16; First posted 2020-12-02 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Endometriosis; Pain
MeSH Terms: conditions — Endometriosis; Pain

STUDY DESIGN:
Intervention Model Description: Randomized, comparative, open-label, controlled interventional pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endocare treatment (Experimental): Patients will receive the treatment on a dedicated virtual reality headset to display the Endocare® application, with high quality headphones
  Interventions: Device: Virtual reality
- Digital control treatment (Active Comparator): Patients will receive the digital control on a dedicated tablet to display the digital control, with high quality headphones
  Interventions: Device: Digital control

INTERVENTIONS:
Device: Virtual reality — 20 minutes treatment in virtual reality
  Arms: Endocare treatment
Device: Digital control — 20 minutes digital control movie on tablet without virtual reality
  Arms: Digital control treatment

SUMMARY:
Endocare® treatment is a stand-alone software medical device, which is composed of a mobile application and an accessory VR headset, intended to mitigate the pain for patients prone to endometriosis.

DETAILED DESCRIPTION:
Endocare® treatment is a stand-alone software medical device, which is composed of a mobile application and an accessory VR headset, intended to mitigate the pain for patients prone to endometriosis.

Mitigation of pain is realized through sequences of treatments via audio and visual stimulations.

The Endocare® treatment's main functionality, which addressed the intended purpose, is conducting sequences for treatment to mitigate the pain sensed by the patient.

The software will allow mitigating the sensed pain through 3D Virtual Reality via sequences of environments. The software will emit through sequences of 3D environments, auditory and visual stimulations.

The medical device is a CE marked Class I device. Women suffering from endometriosis present recurrent pelvic pain impairing their quality of life. The endometriosis-related pain has pejorative repercussions on sexual, family and professional life. Currently, the physician armamentarium is limited to analgesics and non-steroid anti-inflammatory drugs to treat endometriosis-related pain. Endocare® treatment intends to relieve pain thanks to its action on central nervous system. This study will describe the evolution of pain in patients experiencing endometriosis-related pain after a single treatment of Endocare® or a digital control.

The use of a digital control as a comparator is the only way to show a specific effect of the Endocare® treatment. Therefore, a digital control displaying visual and auditive sequences with no expected effect will be used for the study. This digital control, for which only a placebo effect may occur, will be displayed on a tablet instead of VR (Colloca et al., 2020).

The main analysis will be performed on an intent-to-treat basis. The statistical analysis will be performed using the SAS 9.4 (or higher) software (SAS Institute, Cary, NC, USA).

Continuous variables will be described by the number of observations, mean, standard deviation, minimum, maximum and median. Categorical variables will be described by the number and percentage of each modality. Percentages will be calculated on the number of observed data.

ELIGIBILITY:
Inclusion Criteria:

* Woman ≥ 18 years old
* With a diagnosis of endometriosis
* Willing to participate in the study and having signed the informed consent form
* Suffering from a moderate-to-severe endometriosis-related pain ≥ 4 on numerical rating scale (NRS) at the time of inclusion

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Woman having consumed painkillers within 8h prior inclusion
* Woman participating in an interventional study or having participated in an interventional study within the 30 days before enrolment
* Contraindication to Endocare® or digital control: patients with severe visual, hearing and/or cognitive impairments, patients with colour blindness, patients who are photo-sensitive or suffering from epilepsy or motion sickness
* Woman being an employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as family members of the employees or the investigator

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2020-12-03 (Actual); Primary Completion 2021-05-18 (Actual); Study Completion 2021-05-18 (Actual)

PRIMARY OUTCOMES:
Mean pain intensity 60 minutes after the beginning of treatment | 60 minutes after treatment
  Pain assessment evaluated with numerical rating scale (NRS):
  Pain assessed by 11-point numerical rating scale (NRS):
  0=no pain; 10=unbearable pain

SECONDARY OUTCOMES:
Evaluate the pain evolution after Endocare® compared to the digital control | baseline (before treatment), 15 minutes, 30 minutes, 45 minutes, and 240 minutes after treatment
  Pain assessment evaluated with numerical rating scale (NRS):
  11-point numerical scale (0=no pain; 10=unbearable pain)
Evaluate the pain relief after Endocare ® compared to the digital control | 15 minutes, 30 minutes, 45 minutes, 60 minutes, 240 minutes after treatment
  The time to reach and maintain pain relief as assessed by the pain relief score ≥ 3
  PRS is a 5-point categorical scale (0: no relief, 1: slight relief, 2: moderate relief, 3: lots of relief and 4: complete relief)
  The event will be defined by the first occurrence of PRS ≥ 3
Evaluate the maximum reduction in pain after Endocare® compared to the digital control | 15 minutes, 30 minutes, 45 minutes, 60 minutes, 240 minutes after treatment
  The time to reach and maintain pain reduction ≥30% and ≥50% evaluated with NRS 11-point numerical scale (0=no pain; 10=unbearable pain)
Describe the women satisfaction toward Endocare® or the digital control | 240 minutes after treatment
  Satisfaction after using Endocare® compared to the digital control, will be self-rated by the patient on a 7-point Likert scale:
  1: extremely dissatisfied, 2: very dissatisfied, 3: rather dissatisfied, 4: neutral, 5: rather satisfied, 6: very satisfied, 7: extremely satisfied
Evaluate the safety of Endocare® or the digital control | through study completion, at 240 minutes after treatment
  Incidence of adverse events (AE)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Merlot, MD, Principal Investigator — Clinique Tivoli Ducos
Locations (1):
- Clinique Tivoli Ducos, Bordeaux, Gironde, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Merlot B, Dispersyn G, Husson Z, Chanavaz-Lacheray I, Dennis T, Greco-Vuilloud J, Fougere M, Potvin S, Cotty-Eslous M, Roman H, Marchand S. Pain Reduction With an Immersive Digital Therapeutic Tool in Women Living With Endometriosis-Related Pelvic Pain: Randomized Controlled Trial. J Med Internet Res. 2022 Sep 21;24(9):e39531. doi: 10.2196/39531. PMID 36129733